CLINICAL TRIAL: NCT03872700
Title: A Randomized Trial of Intranasal Fentanyl Versus Placebo as an Adjunct to Lidocaine Infiltration in Adults Undergoing Abscess Incision and Drainage in the Emergency
Brief Title: Intranasal Fentanyl as an Adjunct to Lidocaine Infiltration in Adults Undergoing Abscess Incision and Drainage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-9925
Record Dates: First submitted 2019-01-24; First posted 2019-03-13 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Abscess
MeSH Terms: conditions — Abscess

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intranasal fentanyl (Experimental): 2 mcg/kg INF, administered via intranasal route by atomizer syringe
  Interventions: Drug: Intranasal fentanyl
- Placebo (Experimental): 0.04ml/kg of sterile water, administered via intranasal route by atomizer syringe
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal fentanyl — Fentanyl Citrate
  Arms: Intranasal fentanyl
Drug: Placebo — Sterile Water Up to 5Cc
  Arms: Placebo

SUMMARY:
This randomized clinical trial aims to compare the analgesic efficacy of intranasal fentanyl to placebo as analgesic adjunct to conventional local anesthesia for the treatment of pain of the overall procedure in adult patients undergoing lidocaine infiltration and subsequent abscess incision and drainage in the Emergency Department (ED).

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the ED for an abscess requiring incision and drainage
* ED attending physician's judgment that the patient has capacity to provide informed consent.
* Patients must be able to understand English or Spanish.

Exclusion Criteria:

* Use of opioids or tramadol within past 7 days.
* Prior adverse reaction or allergy to opioids.
* Patients who are pregnant
* Patients weight > 100kg
* Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in modulation of pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
* Medical condition that might affect metabolism or opioid analgesics such as cirrhosis (Child Pugh A or worse) or kidney impairment (CKD 3 or worse)
* Chronic malnutrition, severe hypovolemia (dehydration of blood loss) or hepatic disease
* Alcohol intoxication: history of alcoholism or the presence of alcohol intoxication as judged by the treating physician may alter pain perception and has previously increased adverse events.
* SBP <100 mmHg: Opioids can produce peripheral vasodilation causing orthostasis.
* HR < 60/min: Opioids can cause bradycardia.
* Oxygen saturation < 95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
* Use of MAO inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
* Patients using transdermal pain patches or oral opioid use > 10 days in the prior month: frequent opioid use may influence both the amount of pain patients report as well as the level of relief they obtain from other treatments.
* Patients with a history of traumatic brain injury, seizures or hallucinations
* Patients with anatomical anomalies or medical conditions precluding intranasal administration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halvorson GD, Halvorson JE, Iserson KV. Abscess incision and drainage in the emergency department--Part I. J Emerg Med. 1985;3(3):227-32. doi: 10.1016/0736-4679(85)90077-0. PMID 4093575
- [Background] Chudnofsky CR, Wright SW, Dronen SC, Borron SW, Wright MB. The safety of fentanyl use in the emergency department. Ann Emerg Med. 1989 Jun;18(6):635-9. doi: 10.1016/s0196-0644(89)80517-7. PMID 2729688
- [Background] Qualls ML, Mooney MM, Camargo CA Jr, Zucconi T, Hooper DC, Pallin DJ. Emergency department visit rates for abscess versus other skin infections during the emergence of community-associated methicillin-resistant Staphylococcus aureus, 1997-2007. Clin Infect Dis. 2012 Jul;55(1):103-5. doi: 10.1093/cid/cis342. Epub 2012 Mar 28. PMID 22460965
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Brown JC, Klein EJ, Lewis CW, Johnston BD, Cummings P. Emergency department analgesia for fracture pain. Ann Emerg Med. 2003 Aug;42(2):197-205. doi: 10.1067/mem.2003.275. PMID 12883507
- [Background] Lewis LM, Lasater LC, Brooks CB. Are emergency physicians too stingy with analgesics? South Med J. 1994 Jan;87(1):7-9. doi: 10.1097/00007611-199401000-00002. PMID 8284721
- [Background] Schmitz G, Goodwin T, Singer A, Kessler CS, Bruner D, Larrabee H, May L, Luber SD, Williams J, Bhat R. The treatment of cutaneous abscesses: comparison of emergency medicine providers' practice patterns. West J Emerg Med. 2013 Feb;14(1):23-8. doi: 10.5811/westjem.2011.9.6856. PMID 23447753
- [Background] Bourne CL, Brewer KL, House J. Injectable lidocaine provides similar analgesia compared to transdermal lidocaine/tetracaine patch for the incision and drainage of skin abscesses: a randomized, controlled trial. J Emerg Med. 2014 Sep;47(3):367-71. doi: 10.1016/j.jemermed.2013.11.126. Epub 2014 May 14. PMID 24835497
- [Background] Chang AK, Bijur PE, Baccelieri A, Gallagher EJ. Efficacy and safety profile of a single dose of hydromorphone compared with morphine in older adults with acute, severe pain: a prospective, randomized, double-blind clinical trial. Am J Geriatr Pharmacother. 2009 Feb;7(1):1-10. doi: 10.1016/j.amjopharm.2009.02.002. PMID 19281935
- [Background] Chang AK, Bijur PE, Davitt M, Gallagher EJ. Randomized clinical trial of an intravenous hydromorphone titration protocol versus usual care for management of acute pain in older emergency department patients. Drugs Aging. 2013 Sep;30(9):747-54. doi: 10.1007/s40266-013-0103-y. PMID 23846749
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- [Background] McNamara RM, Rousseau E, Sanders AB. Geriatric emergency medicine: a survey of practicing emergency physicians. Ann Emerg Med. 1992 Jul;21(7):796-801. doi: 10.1016/s0196-0644(05)81024-8. PMID 1610035
- [Background] Potter M, Schafer S, Gonzalez-Mendez E, Gjeltema K, Lopez A, Wu J, Pedrin R, Cozen M, Wilson R, Thom D, Croughan-Minihane M. Opioids for chronic nonmalignant pain. Attitudes and practices of primary care physicians in the UCSF/Stanford Collaborative Research Network. University of California, San Francisco. J Fam Pract. 2001 Feb;50(2):145-51. PMID 11219563
- [Background] Petrack EM, Christopher NC, Kriwinsky J. Pain management in the emergency department: patterns of analgesic utilization. Pediatrics. 1997 May;99(5):711-4. doi: 10.1542/peds.99.5.711. PMID 9113948
- [Background] Borland M, Milsom S, Esson A. Equivalency of two concentrations of fentanyl administered by the intranasal route for acute analgesia in children in a paediatric emergency department: a randomized controlled trial. Emerg Med Australas. 2011 Apr;23(2):202-8. doi: 10.1111/j.1742-6723.2011.01391.x. Epub 2011 Feb 8. PMID 21489168
- [Background] Panagiotou I, Mystakidou K. Intranasal fentanyl: from pharmacokinetics and bioavailability to current treatment applications. Expert Rev Anticancer Ther. 2010 Jul;10(7):1009-21. doi: 10.1586/era.10.77. PMID 20645689
- [Background] Paech MJ, Lim CB, Banks SL, Rucklidge MW, Doherty DA. A new formulation of nasal fentanyl spray for postoperative analgesia: a pilot study. Anaesthesia. 2003 Aug;58(8):740-4. doi: 10.1046/j.1365-2044.2003.03286.x. PMID 12859464
- [Background] Veldhorst-Janssen NM, Fiddelers AA, van der Kuy PH, Kessels AG, Theunissen HM, van der Hulst RR, Neef C, Marcus MA. Pharmacokinetics, analgesic effect, and tolerability of a single preprocedural dose of intranasal fentanyl in patients undergoing drain removal after breast reduction or augmentation surgery: A prospective, randomized, double-blind, placebo-controlled study. Clin Ther. 2010 Jul;32(7):1427-36. doi: 10.1016/j.clinthera.2010.07.001. PMID 20678689
- [Background] Toussaint S, Maidl J, Schwagmeier R, Striebel HW. Patient-controlled intranasal analgesia: effective alternative to intravenous PCA for postoperative pain relief. Can J Anaesth. 2000 Apr;47(4):299-302. doi: 10.1007/BF03020941. PMID 10764171
- [Background] Barrett MJ, Cronin J, Murphy A, McCoy S, Hayden J, an Fhaili S, Grant T, Wakai A, McMahon C, Walsh S, O'Sullivan R. Intranasal fentanyl versus intravenous morphine in the emergency department treatment of severe painful sickle cell crises in children: study protocol for a randomised controlled trial. Trials. 2012 May 30;13:74. doi: 10.1186/1745-6215-13-74. PMID 22647439
- [Background] Sutter ME, Wintemute GJ, Clarke SO, Roche BM, Chenoweth JA, Gutierrez R, Albertson TE. The Changing Use of Intravenous Opioids in an Emergency Department. West J Emerg Med. 2015 Dec;16(7):1079-83. doi: 10.5811/westjem.2015.10.28454. Epub 2015 Dec 14. PMID 26759658
- [Background] Imamoglu M, Aygun A, Bekar O, Erdem E, Cicek M, Tatli O, Karaca Y, Sahin A, Turkmen S, Turedi S. A retrospective analysis of nebulized versus intravenous fentanyl for renal colic. Am J Emerg Med. 2017 May;35(5):757-763. doi: 10.1016/j.ajem.2017.01.026. Epub 2017 Jan 15. PMID 28119014
- [Background] Price DD, Finniss DG, Benedetti F. A comprehensive review of the placebo effect: recent advances and current thought. Annu Rev Psychol. 2008;59:565-90. doi: 10.1146/annurev.psych.59.113006.095941. PMID 17550344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in August 2019, was temporarily suspended from March 2020 through June 2020 due to COVID-19. Enrollment was permanently halted by the data safety monitoring committee in April 2021 due to inadequate accrual. During the 19 months in which the study was open for enrollment, 176 patients were screened for eligibility and 49 patients were enrolled.
Period: Overall Study
Arm/Group | Intranasal Fentanyl | Placebo
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Fentanyl | Placebo | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (11) | 36.8 (10.3) | 36.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain Score at Baseline
Description: Patient reported pain scores at baseline. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale | 8.3 (1.5) | 8.1 (2.9)

2. Primary Outcome: NRS Pain Score After Lidocaine Injection
Description: Patient reported NRS pain scores after Lidocaine injection. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Following Lidocaine injection measured once anytime up to 12 minutes after intranasal administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale | 8.4 (2.7) | 8.0 (2.2)

3. Primary Outcome: NRS Pain Score Following Incision
Description: Patient reported NRS pain scores following Incision. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Measured once anytime up to 60 minutes following intranasal administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale | 3.9 (3.6) | 3.9 (3.8)

4. Primary Outcome: NRS Pain Score After Blunt Dissection
Description: Patient reported NRS pain scores after Blunt Dissection. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Measured once anytime up to 60 minutes following intranasal administration
Population: Only 22 patients in each arm received Blunt Dissection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale | 4.1 (4.0) | 4.4 (3.8)

5. Primary Outcome: NRS Pain Score After Irrigation
Description: Patient reported NRS pain scores after Irrigation. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Measured once anytime up to 60 minutes following intranasal administration
Population: Only 23 patients in the Intranasal Fentanyl arm and only 21 patients in the Placebo arm received Irrigation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 23 | 21
score on a scale | 3.4 (3.8) | 2.6 (3.4)

6. Primary Outcome: NRS Pain Score After Packing of Abscess
Description: Patient reported pain after Packing of abscess. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Measured once at the time of completion of application of the bandage, up to 60 minutes following intranasal administration
Population: Only 23 patients in the Intranasal Fentanyl arm and only 22 patients in the Placebo arm received Packing of abscess
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 23 | 22
score on a scale | 4.5 (3.9) | 3.9 (3.8)

7. Primary Outcome: Numerical Rating Scale (NRS) Pain Score for Overall Procedure
Description: Patient reported pain scores for overall Procedure assessed immediately after placement of dressing at the end of procedure. The NRS for pain is a reliable and validated measure of pain intensity ranging from 0 - no pain, to 10 - worst pain imaginable.
Time Frame: Measured once following placement of dressing at completion of procedure, up to 60 minutes following intranasal administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale | 6.2 (3.3) | 7.0 (3.2)

8. Secondary Outcome: Patient Satisfaction With Analgesia
Description: Patient reported outcomes were measured and reported using the Descriptive Scale below:
  Descriptive Scale: satisfied with analgesia, neutral, not satisfied with analgesia
  *This is a non-numerical scale with 3 outcome response options as listed above. Satisfied is rated higher than neutral which is, in turn, rated higher than not satisfied.
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 24 | 25
Participants
  Not Satisfied with Analgesia | 1 | 4
  Neutral (neither satisfied nor dis-satisifed) | 9 | 13
  Satisfied with Analgesia | 14 | 8

9. Secondary Outcome: Health Care Providers Reported Perception of Study Medication Compared to Usual Care
Description: Provider perception of better, same or worse treatment compared to usual care
  Descriptive Scale: better, same, worse
  *This is a non-numerical scale with 3 outcome response options as listed above. Better is rated higher than same which is, in turn, rated higher than worse.
Time Frame: 120 minutes
Population: This study was formally completed as per Albert Einstein College of Medicine IRB records. Data was not collected for the Health care providers reported perception of study medication compared to usual care' outcome and as such an assessment of whether study medication provided a better, worse, or similar outcome as compared to usual care, from a provider perspective, was unable to be made
Arm/Group | Intranasal Fentanyl | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 60 minutes following initiation of treatment administration
Description: Subjects were assessed for medication-related adverse effects by being queried for the onset of any new symptoms that began following receipt of the study medication. Affirmative responses were followed by an open-ended question eliciting details. All adverse events, including medication-related and non medication-related adverse events are summarized in the Adverse Events module.
Arm/Group | Intranasal Fentanyl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 3/24 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Fentanyl (N=24) | Placebo (N=25)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Drowsiness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sadness (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03872700/Prot_SAP_002.pdf
  • Informed Consent Form (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03872700/ICF_001.pdf